CLINICAL TRIAL: NCT03286478
Title: A Cluster Randomised Controlled Trial of Three School-based Body Image Interventions Delivered by Teachers
Brief Title: A Trial of Three School-based Body Image Interventions Delivered by Teachers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of the West of England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SFS-16-001
Record Dates: First submitted 2017-09-08; First posted 2017-09-18 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Body Image
Keywords: body image; school; adolescence; intervention; task-shifting
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Parallel 4-arm cluster randomised controlled trial.
Masking Description: Masking not possible within design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness (Experimental): Mindfulness-based body image intervention
  Interventions: Behavioral: Mindfulness
- Dissonance (Experimental): Cognitive dissonance-based body image intervention
  Interventions: Behavioral: Dissonance
- Confident Me (Experimental): Dove Confident Me body image intervention
  Interventions: Behavioral: Dove Confident Me
- Control (No Intervention): Classes as usual, assessment-only control group.

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness-based body image intervention to be delivered 1 lesson per week for 5 weeks (5 x 45 minute lessons), by trained school teachers.
  Arms: Mindfulness
Behavioral: Dissonance — Dissonance-based body image intervention to be delivered 1 lesson per week for 5 weeks (5 x 45 minute lessons), by trained school teachers.
  Arms: Dissonance
Behavioral: Dove Confident Me — Dove Confident Me body image intervention to be delivered 1 lesson per week for 5 weeks (5 x 45 minute lessons), by trained school teachers.
  Arms: Confident Me

SUMMARY:
Body image is one of the leading concerns for young people. Such concerns can have serious health consequences, including unhealthy weight control and exercise behaviours, depression, smoking, low self-esteem and misusing drugs and alcohol. Leading and emerging approaches for improving body image are effective among older adolescent females, and when delivered by expert providers (e.g., psychologists). However, there is a need for body image programmes that include males and so can be delivered in co-educational settings, and can be delivered by non-expert providers (e.g., teachers within schools) to facilitate cost-effective and ongoing use.

This project will evaluate three classroom-based programmes for improving young people's body image, delivered by class teachers to girls and boys aged 13-14 years in secondary schools. Two programmes are based on leading (cognitive dissonance) and emerging (mindfulness) approaches for improving body image, but which have not been previously evaluated with both boys and girls and when delivered by teachers. The third programme has previously demonstrated effectiveness in improving body image when delivered by teachers to boys and girls in the classroom setting, and therefore will provide a useful comparison to benchmark these programmes.

To assess the impact of each programme, the current study will compare the body image and well-being of students who take part in each programme to students who take part in an alternative programme, and those who do not take part in any programme (classes as usual), over a 6-month period. The investigators will also assess the extent to which gender and pre-existing levels of body image concerns impacts the benefit received from taking part in the lessons. To undertake this project, the investigators will recruit students and teachers from 24 schools in Bristol and surrounding areas in the South West of England. Students will complete questionnaire assessments of body image and well-being before and after the 5-week programme period, and again 6 months later to assess longer-term benefits. The investigators will also gain in-depth feedback from students and teachers via focus groups and interviews, in order to inform future improvement of the programmes for wider implementation.

Therefore, this trial will assess whether the two newly adapted programmes result in improved body image compared to those who receive their classes as usual, and compared to an existing teacher-led programme.

DETAILED DESCRIPTION:
Background:

Body image is recognised as an important public health issue by governments, policy-makers, and health professionals. Poor body image is associated with engagement in unhealthy weight loss behaviours, depression, reduced academic performance, and has been established as an important risk factor in the development eating disorders. Within Western societies, poor body image is also common, with an estimated 25-61% of adolescent girls and boys being dissatisfied with their appearance. This underlines the importance of prevention and early intervention. As such, researchers, governments and health professionals are increasingly seeking effective evidence-based body image interventions that can be disseminated to the public, in a bid to reduce body image concerns and other adverse negative health related effects such as eating disorders. However, widespread dissemination of these programmes remains a challenge due to the difficulty of reaching individuals at risk, the traditional focus on females only, and the reliance on expert intervention facilitators.

Although it can be difficult reaching those at risk with individual targeted prevention programs, school-based interventions provide a useful opportunity to reach large and diverse groups of children and young people, crossing all levels of risk and gaining access to those who may otherwise not receive necessary intervention. Effective school-based interventions are designed to reduce the presence or influence of risk factors for body image concerns (e.g., internalisation of appearance ideals, appearance pressures from friends, family and the media, appearance-related teasing and bullying, and negative emotions such as depression and anxiety) in an effort to promote healthy body image. Previous school-based work has demonstrated some success in reducing body concerns at the conclusion of program implementation and over meaningful follow-up periods, with evidence showing media literacy and cognitive dissonance approaches to be useful in this context. However, there is still room for improvement in the magnitude of effects for universal programmes, and the majority are still targeted at girls and led by expert facilitators. Consequently, further evaluation of different approaches in this setting is required.

In addition, another factor which is still rather mixed within the literature, and has an impact on how universal programmes are delivered, is regarding the use of expert-led versus teacher-led interventions. Previous reviews have shown that programs are more effective when facilitated by dedicated expert interventionists. However, evidence from previous studies conducted by the investigators supports the notion that teachers can deliver a body image intervention effectively with minimal training. Hence, more research is needed to understand the effectiveness of teacher led interventions further, as successful task-shifting to non-expert providers has been identified as an important goal for disseminating mental health interventions at scale.

Therefore, the aim of this research is to evaluate the efficacy and acceptability of adapted interventions based on mindfulness and cognitive dissonance, respectively, for delivery to adolescent girls and boys (aged 13-14 years) by trained teachers. They will be compared against an existing universal intervention with support for teacher-led delivery and a class-as-usual control group.

Design:

This study will be a parallel 4-arm cluster randomised controlled trial. Schools will be randomly allocated to receive either the cognitive dissonance, mindfulness, or Dove Confident Me interventions, or classes-as-usual (control). The intervention duration is the same for all experimental conditions, and students will be assessed on body image and related outcomes at baseline, post-intervention, and 6-month follow-up (with 12-month planned pending further funding).

Participants, recruitment, and allocation:

Sample size for our repeated measures design was determined a priori. Assuming a small effect size of Cohen's d = .2 based on previous research of teacher-led programmes, a medium intra-individual correlation between repeated measures of .5, and setting power at .80, the sample size required to detect significance at the 5% level under individual randomisation was 294 students per arm. Applying an inflation factor to account for school level clustering based on a small intraclass correlation coefficient (ICC) of .01 (informed by previous studies), increased this requirement to 585 students per arm. Based on an average of 100 students from Grade 9 classes per school, the investigators aim to recruit 6 schools per arm. Thus the investigators aim to recruit 24 secondary schools in total (N = 2400 students) from Bristol and surrounding areas (UK).

Schools will be initially invited to take part via email and phone, and via involvement in a wider programme aimed at facilitating greater participation in higher education run by the Widening Participation team at the host institution. Allocation will be undertaken using restricted randomisation based on minimisation in order to achieve balance in each of the arms with regard to key school characteristics (geographical region, socioeconomic status, proportion of students learning English as a second language). This is the recommended approach for cluster randomised controlled trials (RCTs) that recruit and allocate sequentially, and will be implemented using freely available computer software (Minim).

Interventions:

Dove Confident Me

Dove Confident Me represents an existing school-based intervention that targets multiple risk factors for body dissatisfaction, addressing the nature and source of societal appearance ideals, media literacy, appearance-related social comparisons, appearance-related conversations and teasing, and encouraging 'body activism' to challenge appearance pressures. It consists of five 45-minute interactive lessons, designed to be delivered by teachers in school classrooms. The intervention was an adaptation of an existing evidence-based expert-led programme, Happy Being Me. Standardised materials include a detailed lesson plan for teachers, PowerPoint slides, video clips, and student activity sheets. Intervention materials are freely available online in five languages (selfesteem.dove.com).

Cognitive dissonance

Cognitive dissonance is conceptualised as the psychological discomfort stemming from conflicting cognitions and behaviours. Inducing such a state can be used to shift targeted attitudes and behaviours, as individuals are motivated to do so order regain equilibrium. In the context of body image and eating disorder prevention, dissonance-based interventions (DBIs) encourage a voluntary counter-attitudinal stance against socially prescribed appearance ideals in order to produce a conflict with, and therefore reduce, internalization of such ideals and their consequences. An existing school-based dissonance intervention which was previously tested among early adolescent girls with psychologist delivery has been adapted for delivery to mixed-gender adolescents by trained teachers. It has been designed to follow the same format and length as Dove Confident Me, and therefore consists of 5 x 45minute lessons, with detailed lesson plans for teachers, accompanying Powerpoint presentations and student activity sheets.

Mindfulness

Mindfulness refers to the awareness and acceptance of present-moment experience. As a psychological technique, it is growing in support for treating a range of mental health concerns. Mindfulness based interventions (MBI) are the next potential alternative to cognitive dissonance interventions (CDI) as they represent a potentially useful strategy for promoting positive body image. In this context, MBIs aim to both increase the capacity to refrain from automatic responses when confronted with appearance ideals and related sociocultural pressures, and reduce the intensity and impact of negative experiences if and when they do occur. An existing school-based mindfulness intervention which the investigators have previously tested among older adolescent girls with psychologist delivery has been adapted for delivery to adolescent girls and boys by trained teachers. It has been designed to follow the same format and length as Dove Confident Me, and therefore consists of 5 x 45minute lessons, with detailed lesson plans for teachers, accompanying Powerpoint presentations and student activity sheets.

Procedure Informed active consent will be obtained from school senior management (during recruitment), informed assent from parents (prior to baseline assessment), and informed consent from students (at baseline assessment). Prior to lesson delivery, school teachers will be trained in their allocated intervention by expert body image researchers (2 x 1.5hr sessions), and will be provided with all teaching materials necessary for delivering the interventions. Students will complete questionnaires under standardised conditions supervised by their teachers and trained research staff. Approximately one week following baseline questionnaires, intervention schools will deliver their allocated intervention, facilitated by schoolteachers to whole classes (one lesson per week over five weeks), with a ratio of one teacher to 20-30 students. All lessons will be audio-recorded and a selection of lessons will be observed live by trained research staff, for the purposes of assessing fidelity to the intervention manuals. Teachers and selected students will take part in focus group interviews following completion of the lessons, in order to obtain qualitative feedback. Students in control schools will take part part in their usual scheduled lessons. All students will then complete follow-up questionnaires at post-intervention (within one week of final lesson), and 6-month follow-up. Blinding of students, teachers, and researchers is not possible due to the nature of the interventions. However, risk of bias from teachers and researchers is minimised due to anonymous self-report assessments. Risk of contagion is also minimised by randomising at the school level. Participating schools will receive a £200 honorarium upon project completion. This project has received ethical approval from the University of the West of England's Faculty Research Ethics Committee (HAS.16.09.016).

Statistical analysis plan:

Multiple imputation will be used to handle missing data. Analysis of intervention effects will be conducted using an intent-to-treat approach, with a sensitivity analysis conducted depending on the extent of missing data. Multilevel mixed models will be used to compare groups at post-intervention and 6-month follow-up on primary and secondary outcomes, accounting for the clustered nature of the design (repeated measures within students, within classes, within schools). Baseline levels of outcomes, as well as demographic and school characteristics will be used as covariates in order to increase precision of effects. Follow-up analysis will investigate moderation with respect to gender and baseline body image concerns, and will be conducted by including interactional terms in the statistical models. Subsequent mediational analyses following recommendations by Kraemer will investigate hypothesised mechanisms of change in each of the trial arms. An analysis of cost-effectiveness will also be undertaken, comparing relative effectiveness across interventions.

ELIGIBILITY:
Inclusion Criteria (school):

* Co-educational secondary school
* Available to include Year 9 classes in the study

Exclusion Criteria (school):

* Single-sex schools
* Not available to include Year 9 classes in the study

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline body esteem over time | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of global body image using the Body Esteem Scale for Adolescents and Adults, 5-point Likert-type scale, 18 items
Change in baseline body satisfaction over time | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of body dissatisfaction with specific body parts using the Body Satisfaction (Project Eat III), 5 point Likert-type scale, 14 items
Change in eating pathology over time | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of eating disorder psychopathology using Eating Disorder Examination-Questionnaire-Short, 4 point Likert-type scale, 12 items

SECONDARY OUTCOMES:
Sociocultural Attitudes Towards Appearance Questionnaire-3 (Internalisation subscale) | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of internalisation of appearance ideals (proposed mediator of The Body Project), 5 point Likert-type scale, 9 items
Comprehensive Inventory of Mindfulness Experiences-Adolescents | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of mindfulness (proposed mediators of the Mindfulness Mode), 4 point Likert-type scale, 25 items
Media Literacy Scale - Commercially generated and Peer-generated subscales | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of media literacy (proposed mediator of Dove Confident Me), 5 point Likert-type scale, 20 items
Positive and Negative Affect Scale for Children | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of positive and negative emotional states, 5 point Likert-type scale, 10 items
Life Engagement Scale | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of the psychosocial impact of body image concerns, 4 point Likert-type scale, 10 items
Depression, Anxiety and Stress Scales-21 | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of mental well-being (depression, anxiety and stress), 4 point Likert-type scale, 21 items
EuroQol health related quality of life - Youth (EQ-5D-Y) | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Assessment of overall health status in order to calculate Quality Adjusted Life Years, 3-point scale, 5 items, plus a single 100 point item
Academic achievement | Baseline, post-intervention (6-week), 6-month, 12-month (pending further funding)
  Self-report two most commonly received school grades (A,B,C,D,E,F, Incomplete)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Atkinson, PhD, Principal Investigator — University of the West of England; Phillippa C Diedrichs, PhD, Principal Investigator — University of the West of England
Locations (1):
- University of the West of England, Bristol, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diedrichs PC, Atkinson MJ, Steer RJ, Garbett KM, Rumsey N, Halliwell E. Effectiveness of a brief school-based body image intervention 'Dove Confident Me: Single Session' when delivered by teachers and researchers: Results from a cluster randomised controlled trial. Behav Res Ther. 2015 Nov;74:94-104. doi: 10.1016/j.brat.2015.09.004. Epub 2015 Sep 30. PMID 26469131
- [Background] Atkinson MJ, Wade TD. Mindfulness-based prevention for eating disorders: A school-based cluster randomized controlled study. Int J Eat Disord. 2015 Nov;48(7):1024-37. doi: 10.1002/eat.22416. Epub 2015 Jun 6. PMID 26052831
- [Background] Halliwell E, Yager Z, Paraskeva N, Diedrichs PC, Smith H, White P. Body Image in Primary Schools: A pilot evaluation of a primary school intervention program designed by teachers to improve children's body satisfaction. Body Image. 2016 Dec;19:133-141. doi: 10.1016/j.bodyim.2016.09.002. Epub 2016 Sep 28. PMID 27693763
- [Background] Yager Z, Diedrichs PC, Ricciardelli LA, Halliwell E. What works in secondary schools? A systematic review of classroom-based body image programs. Body Image. 2013 Jun;10(3):271-81. doi: 10.1016/j.bodyim.2013.04.001. Epub 2013 May 14. PMID 23683611
- [Background] Halliwell E, Diedrichs PC. Testing a dissonance body image intervention among young girls. Health Psychol. 2014 Feb;33(2):201-4. doi: 10.1037/a0032585. Epub 2013 May 13. PMID 23668845
- [Background] Bird EL, Halliwell E, Diedrichs PC, Harcourt D. Happy Being Me in the UK: a controlled evaluation of a school-based body image intervention with pre-adolescent children. Body Image. 2013 Jun;10(3):326-34. doi: 10.1016/j.bodyim.2013.02.008. Epub 2013 Apr 3. PMID 23562583
- [Background] Stice E, Shaw H, Becker CB, Rohde P. Dissonance-based Interventions for the prevention of eating disorders: using persuasion principles to promote health. Prev Sci. 2008 Jun;9(2):114-28. doi: 10.1007/s11121-008-0093-x. Epub 2008 May 28. PMID 18506621
- [Background] Al Sabbah H, Vereecken CA, Elgar FJ, Nansel T, Aasvee K, Abdeen Z, Ojala K, Ahluwalia N, Maes L. Body weight dissatisfaction and communication with parents among adolescents in 24 countries: international cross-sectional survey. BMC Public Health. 2009 Feb 6;9:52. doi: 10.1186/1471-2458-9-52. PMID 19200369
- [Background] Xie B, Unger JB, Gallaher P, Johnson CA, Wu Q, Chou CP. Overweight, body image, and depression in Asian and Hispanic adolescents. Am J Health Behav. 2010 Jul-Aug;34(4):476-88. doi: 10.5993/ajhb.34.4.9. PMID 20218759
- [Background] Neumark-Sztainer D, Paxton SJ, Hannan PJ, Haines J, Story M. Does body satisfaction matter? Five-year longitudinal associations between body satisfaction and health behaviors in adolescent females and males. J Adolesc Health. 2006 Aug;39(2):244-51. doi: 10.1016/j.jadohealth.2005.12.001. PMID 16857537
- [Background] Halliwell E, Jarman H, McNamara A, Risdon H, Jankowski G. Dissemination of evidence-based body image interventions: A pilot study into the effectiveness of using undergraduate students as interventionists in secondary schools. Body Image. 2015 Jun;14:1-4. doi: 10.1016/j.bodyim.2015.02.002. Epub 2015 Mar 21. PMID 25805217
- [Background] Atkinson MJ, Wade TD. Enhancing dissemination in selective eating disorders prevention: an investigation of voluntary participation among female university students. Behav Res Ther. 2013 Dec;51(12):806-16. doi: 10.1016/j.brat.2013.09.012. Epub 2013 Oct 9. PMID 24140874
- [Background] Wilksch SM, Paxton SJ, Byrne SM, Austin SB, McLean SA, Thompson KM, Dorairaj K, Wade TD. Prevention Across the Spectrum: a randomized controlled trial of three programs to reduce risk factors for both eating disorders and obesity. Psychol Med. 2015 Jul;45(9):1811-23. doi: 10.1017/S003329171400289X. Epub 2014 Dec 19. PMID 25524249
- [Background] Fairburn CG, Patel V. The global dissemination of psychological treatments: a road map for research and practice. Am J Psychiatry. 2014 May;171(5):495-8. doi: 10.1176/appi.ajp.2013.13111546. No abstract available. PMID 24788281
- [Background] Sharpe H, Schober I, Treasure J, Schmidt U. Feasibility, acceptability and efficacy of a school-based prevention programme for eating disorders: cluster randomised controlled trial. Br J Psychiatry. 2013 Dec;203(6):428-35. doi: 10.1192/bjp.bp.113.128199. Epub 2013 Oct 10. PMID 24115345
- [Background] Ivers NM, Halperin IJ, Barnsley J, Grimshaw JM, Shah BR, Tu K, Upshur R, Zwarenstein M. Allocation techniques for balance at baseline in cluster randomized trials: a methodological review. Trials. 2012 Aug 1;13:120. doi: 10.1186/1745-6215-13-120. PMID 22853820
- [Background] Richardson SM, Paxton SJ. An evaluation of a body image intervention based on risk factors for body dissatisfaction: a controlled study with adolescent girls. Int J Eat Disord. 2010 Mar;43(2):112-22. doi: 10.1002/eat.20682. PMID 19350648
- [Background] Kraemer HC, Wilson GT, Fairburn CG, Agras WS. Mediators and moderators of treatment effects in randomized clinical trials. Arch Gen Psychiatry. 2002 Oct;59(10):877-83. doi: 10.1001/archpsyc.59.10.877. PMID 12365874